CLINICAL TRIAL: NCT01886716
Title: Cognitive Bias Modification: A Novel Intervention for Alcohol Dependence and Social Anxiety
Brief Title: Retraining Attention to Treat Alcohol Dependence and Social Anxiety
Acronym: AMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Miami University (Other); Brown University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Joshua Magee, Assistant Research Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21AA021151 (NIH); 1R21AA021151 (NIH)
Record Dates: First submitted 2013-06-17; First posted 2013-06-26 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Alcohol Drinking; Anxiety Disorders
Keywords: Alcohol Abuse; Alcohol Dependence; Alcohol Drinking; Social Anxiety; Social Phobia; Anxiety Disorders
MeSH Terms: conditions — Alcohol Drinking; Anxiety Disorders; Alcoholism; Phobia, Social | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Anxiety Attention Training only (Experimental): Participants will receive Anxiety Attention Training and placebo Alcohol training.
  Interventions: Behavioral: Anxiety Attention Training
- Alcohol Attention Training only (Experimental): Participants will receive Alcohol Attention Training and placebo Anxiety training.
  Interventions: Behavioral: Alcohol Attention Training
- Anxiety + Alcohol Attention Training (Experimental): Participants will receive both Anxiety Attention Training and Alcohol Attention Training.
  Interventions: Behavioral: Anxiety Attention Training; Behavioral: Alcohol Attention Training
- Control Training (Placebo Comparator): Participants will receive placebo Anxiety Training and placebo Alcohol training.
  Interventions: Behavioral: Control Training

INTERVENTIONS:
Behavioral: Anxiety Attention Training — Anxiety Attention Training will preferentially direct participants' attention away from reminders of anxiety.
  Arms: Anxiety + Alcohol Attention Training; Anxiety Attention Training only
Behavioral: Alcohol Attention Training — Alcohol Attention Training will preferentially direct participants' attention away from reminders of alcohol.
  Arms: Alcohol Attention Training only; Anxiety + Alcohol Attention Training
Behavioral: Control Training — Placebo Anxiety Training and Placebo Alcohol Training will not preferentially direct participants' attention away from reminders of anxiety or alcohol.
  Arms: Control Training

SUMMARY:
The purpose of this research is to test a computerized intervention for people with co-occurring social anxiety and alcohol dependence. The intervention seeks to reduce symptoms by shifting attention away from alcohol-relevant and/or socially threatening cues. The investigators expect that participants receiving alcohol or anxiety training will experience reductions in those specific symptoms compared to participants in a control condition. The investigators also expect that participants receiving combined alcohol and anxiety training will show the largest reductions in alcohol and anxiety symptoms, relative to participants in any other condition.

DETAILED DESCRIPTION:
Alcohol Use Disorders (AUDs) and Social Anxiety Disorder are disabling and chronic conditions. In spite of these common and significantly overlapping problems, insight into the mechanisms linking alcohol dependence and social anxiety symptoms is minimal, and there are not well established treatment guidelines for this population. In this study, the investigators seek to develop a computerized intervention for individuals with symptoms of social anxiety and alcohol dependence. The intervention attempts to reduce symptoms by shifting attention away from alcohol-relevant and/or socially threatening cues. The investigators expect that participants receiving alcohol or anxiety training will experience reductions in those specific symptoms compared to participants in a control condition. The investigators also expect that participants receiving combined alcohol and anxiety training will show the largest reductions in alcohol and anxiety symptoms, relative to participants in any other condition.

ELIGIBILITY:
Inclusion Criteria:

* Current alcohol dependence
* Elevated social anxiety symptoms
* Willingness to consider cutting down on drinking

Exclusion Criteria:

* Current psychosis
* Unmanaged manic symptoms
* Significant cognitive impairment
* Other drug use in past month
* Receiving cognitive behavioral therapy for alcohol use disorder or social anxiety
* Unable to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua C Magee, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Department of Family and Community Medicine, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Random assignment occurred during Week 1, the next visit after the baseline orientation session. Out of 115 participants completing the baseline session, 21 dropped out prior to random assignment. To ensure current symptoms, another 8 were excluded due to baseline reports of no or extremely low alcohol consumption and/or social anxiety, leaving 86.
Period: Week 1
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Started | 24 | 20 | 22 | 20
Completed | 24 | 20 | 20 | 18
Not Completed | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Period: Week 2
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Started | 24 | 20 | 20 | 18
Completed | 21 | 18 | 19 | 15
Not Completed | 3 | 2 | 1 | 3
Not completed — Lost to Follow-up | 3 | 2 | 1 | 3
Period: Week 3
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Started | 21 | 18 | 19 | 15
Completed | 20 | 17 | 19 | 14
Not Completed | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Period: Week 4
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Started | 20 | 17 | 19 | 14
Completed | 20 | 17 | 19 | 14
Not Completed | 0 | 0 | 0 | 0
Period: 1-Week Post Follow-Up
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Started | 20 | 17 | 19 | 14
Completed | 20 | 17 | 19 | 14
Not Completed | 0 | 0 | 0 | 0
Period: 1-Month Post Follow-Up
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Started | 20 | 17 | 19 | 14
Completed | 20 | 17 | 19 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who remained in the study through the initial Week 1 session in which random assignment occurred, as well as who reported current symptoms on alcohol consumption and social anxiety measures at the baseline orientation session (see Pre-Assignment Details and Participant Flow).
Groups:
- Total: Total of all reporting groups
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training | Total
Number analyzed (Participants) | 24 | 20 | 22 | 20 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 19 | 21 | 20 | 84
  >=65 years | 0 | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.50 (10.95) | 47.40 (10.94) | 47.68 (9.83) | 39.70 (10.62) | 44.31 (10.93)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 9 | 7 | 10 | 35
  Male | 15 | 11 | 15 | 10 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 10 | 11 | 10 | 45
  White | 10 | 9 | 9 | 6 | 34
  More than one race | 0 | 0 | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 20 | 22 | 20 | 86

OUTCOME MEASURES:

1. Primary Outcome: Liebowitz Social Anxiety Scale
Description: The experimenter-administered Liebowitz Social Anxiety Scale (Liebowitz, 1987) was the primary measure to assess social anxiety symptoms. This well-validated instrument assesses fear and avoidance across a range of 24 social and performance situations during the course of the previous week. A total LSAS score was computed, ranging from 0 (no fear or avoidance) to 144 (the greatest level of fear and avoidance).
Time Frame: Baseline, weekly throughout the 4-week trial, and in the follow-up sessions (1 week and 1 month follow-ups)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Number analyzed (Participants) | 20 | 17 | 19 | 14
units on a scale | 56.80 (30.82) | 60.94 (27.70) | 52.05 (27.23) | 55.05 (26.08)
Statistical Analysis 1: Comparison: Anxiety Attention Training Only vs Alcohol Attention Training Only vs Anxiety + Alcohol Attention Training vs Control Training; The analyses used multilevel modeling to capture both the trajectories of symptoms within individuals (i.e., level 1) and the hypothesized between-subject moderators of these trajectories, alcohol and anxiety attention training (i.e., level 2) across all 7 time points. Note, although all 4 groups are included in this analysis, this analysis specifically compares anxiety vs. control training; Test type: Superiority or Other; p = .40, Mixed Models Analysis; Slope = -.80, Standard Error of Mean .95 — F(1,517) = .71
Statistical Analysis 2: Comparison: Anxiety Attention Training Only vs Alcohol Attention Training Only vs Anxiety + Alcohol Attention Training vs Control Training; The analyses used multilevel modeling to capture both the trajectories of symptoms within individuals (i.e., level 1) and the hypothesized between-subject moderators of these trajectories, alcohol and anxiety attention training (i.e., level 2) across all 7 time points. Note, although all 4 groups are included in this analysis, this analysis specifically compares alcohol vs. control training; Test type: Superiority or Other; p = .78, Mixed Models Analysis; Slope = .27, Standard Error of Mean .95 — F(1,517) = .08

2. Primary Outcome: The Daily Drinking Questionnaire
Description: The Daily Drinking Questionnaire (Collins, Parks, & Marlatt, 1985) was the primary measure used to assess weekly alcohol consumption. This calendar-based measure was administered by the experimenter once per week to monitor changes in symptoms. The measure assessed the total number of drinks in the past week.
Time Frame: Baseline, weekly throughout the 4-week trial, and in the follow-up sessions (1 week and 1 month follow-ups)
Measure: Mean (Standard Deviation); unit: number of drinks
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Number analyzed (Participants) | 20 | 17 | 19 | 14
number of drinks | 30.25 (39.49) | 22.82 (23.03) | 24.65 (24.93) | 18.48 (24.09)
Statistical Analysis 1: Comparison: Anxiety Attention Training Only vs Alcohol Attention Training Only vs Anxiety + Alcohol Attention Training vs Control Training; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .67, Mixed Models Analysis; Slope = -.03, Standard Error of Mean .07 — F(1,517) = .18
Statistical Analysis 2: Comparison: Anxiety Attention Training Only vs Alcohol Attention Training Only vs Anxiety + Alcohol Attention Training vs Control Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .32, Mixed Models Analysis; Slope = .07, Standard Error of Mean .07 — F(1,517) = 1.01

ADVERSE EVENTS:
Time Frame: Monitoring for adverse events occurred at baseline, weekly throughout the 4-week trial, and in the follow-up sessions (1 week and 1 month follow-ups).
Description: Research assistants completed check-ins for concerns. Two measures were also monitored for significant negative changes,the LSAS and AWSC. Participants scoring ≥9 points above their baseline LSAS score or ≥23 on the AWSC were evaluated by the site principal investigator for the possibility of clinical deterioration and/or symptoms requiring emergency intervention (e.g., suicidal ideation with intent).
Arm/Group | Anxiety Attention Training Only | Alcohol Attention Training Only | Anxiety + Alcohol Attention Training | Control Training
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/24 | 0/20 | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No